CLINICAL TRIAL: NCT00606398
Title: Combined Resection of Intra- and Extra-Hepatic Metastases From Colorectal Cancer: A Phase II Trial
Brief Title: Combined Resection of Colorectal Metastases
Acronym: CRC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Dr. Alice Wei, UHN
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIAW1
Record Dates: First submitted 2008-01-21; First posted 2008-02-04 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: Colorectal Cancer
Keywords: colorectal metastases
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: surgical resection for patients with both intra- and extra-hepatic metastases — Simultaneous resection with R0 intent of intra-abdominal metastases from CRC. For patients with extra-abdominal disease, sequential resection will be permitted

SUMMARY:
This is a Phase II study of combined surgical resection for patients with both intra- and extra-hepatic metastases from colorectal cancer. The primary objective is to determine the two-year disease free survival (DFS) of patients who undergo surgical resection of both intra- and extra-hepatic metastases from colorectal cancer. The secondary objectives are to determine the overall survival rate (OS), patterns of treatment failure, treatment efficacy (R0 resection rate), peri-operative morbidity and mortality rates, health related quality of life, and hospital length of stay.

DETAILED DESCRIPTION:
This phase II clinical study will examine the outcomes of surgical therapy for patients with both intra- and extra-hepatic CRC metastases.

The treatment protocol includes surgical resection of metastases from Colorectal cancer. Multi-modality co-interventions such as chemotherapy (neo-adjuvant, or post-operative), radiofrequency ablation (RFA) and/or portal vein embolization (PVE) will be permitted.

The eligibility criteria include: patients with both intra-hepatic and extra-hepatic metastases from colorectal cancer, the number of extra-hepatic metastases must be three or less on pre-operative imaging, all metastatic deposits must be resectable with R0 intent, there must be no contra-indications to major surgery and an ECOG performance status of 0, 1 or 2.

ELIGIBILITY:
Inclusion Criteria:

* Patients with both intra-hepatic and extra-hepatic metastases from colorectal cancer
* Number of extra-hepatic metastases must be 3 or less on pre-operative imaging
* All metastatic deposits must be resectable with clear margins
* No contra-indications to major surgery
* ECOG performance of 0, 1 or 2
* Age 18 or older
* Pregnant women or women of childbearing potential are eligible if they agree to use 2 methods of effective contraception during treatment protocol
* Written informed consent can be obtained

Exclusion Criteria:

* Colorectal primary in situ
* Four or more extra-hepatic lesions on pre-operative imaging
* Significant medical or psychiatric conditions that preclude major surgery or may interfere with patient compliance
* Patients receiving investigational drugs with unknown surgical risks
* Failure to meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2007-06; Primary Completion 2007-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
two-year disease free survival (DFS) | 2 years

SECONDARY OUTCOMES:
Overall survival rate (OS), patterns of treatment failure, treatment efficacy (R0 resection rate), peri-operative morbidity and mortality rates, health related quality of life, hospital length of stay | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Alice Wei, MD, CM, MSc, FRCSC, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada